CLINICAL TRIAL: NCT06656767
Title: Understanding the Evolution of the Somatic Mutational Landscape in Chronic Liver Disease Across Aetiologies and Disease States
Brief Title: Somatic Mutation in Chronic Liver Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: The Wellcome Sanger Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 346024
Record Dates: First submitted 2024-10-16; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-07

CONDITIONS: Chronic Liver Disease; Somatic Mutation
Keywords: Somatic mutations liver

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Liver tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic Liver Disease: A comprehensive atlas of somatic mutation present in chronic liver disease, spanning disease aetiologies and stages.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This study utilises pre-collected samples only.

SUMMARY:
Deaths from chronic liver disease are rising in the UK and around the world. The leading causes are alcohol-related liver disease, metabolic-dysfunction associated steatotic liver disease (MASLD, formerly known as 'non-alcoholic fatty liver disease') and viral hepatitis. Chronic liver disease puts people at significantly increased risk of liver cancer, which in the UK has a 5 year survival of under 15%. Little is understood about how liver cells acquire genetic changes, called somatic mutations, as they progress from healthy cells, to disease, to cancer development. This study aims to investigate these somatic mutations across different causes of chronic liver disease, and different stages of liver disease. The investigators hope this will help us to understand how different insults to the liver put the liver cells under different pressures, resulting in varying genetic changes. By understanding these changes specific to disease aetiology and stage, novel genetic targets may be identified which assist to focus research in identifying specific prognostic, diagnostic and therapeutic tools in chronic liver disease, and improve outcomes for patients.

Tissue, surplus to clinical requirement, from patients were undergoing liver biopsy, liver resection or liver transplantation (tissue sampling from explanted liver) collected by collaborators at University of Texas Southwestern will undergo genomic sequencing at the Wellcome Sanger Institute.

ELIGIBILITY:
Inclusion Criteria:

Pre-collected cohorts of liver tissue collected from adults (male and female) with consent and ethical approval for use in research.

Exclusion Criteria:

Anything outside of the above including samples other than liver tissue, samples where there is no consent or ethical approval for use in research and/or samples from children.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic liver disease
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-07-07 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Somatic mutations in chronic liver disease | 2 years
  Metrics evaluated include the number of somatic mutations, the spectrum of mutational signatures (encompassing base substitutions, indels, genome rearrangements, and copy number changes), and the size and relatedness of clonal populations within liver tissue samples. These collective analysis of these metrics will aim to identify and quantify variations that may contribute to disease development and progression.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Campbell, Principal Investigator — Wellcome Sanger Institute
Locations (1):
- Wellcome Sanger Institute, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No